CLINICAL TRIAL: NCT07139743
Title: A Single-arm, Open-label, Phase I Study to Determine the Safety, Tolerability, and Preliminary Efficacy of Obe-cel in Participants With Refractory Progressive Forms of Multiple Sclerosis
Brief Title: Obe-cel in Refractory Progressive Forms of Multiple Sclerosis
Acronym: BOBCAT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Autolus Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUTO1-MS1; 2024-519552-93-00 (EU CTIS Number); 1011413 (Other: UK IRAS ID)
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Progressive Multiple Sclerosis
Keywords: Multiple sclerosis; Refractory multiple sclerosis; Progressive multiple sclerosis; Obecabtagene autoleucel; Obe-cel
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Single-arm, single group assignment, open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Obecabtagene autoleucel (obe-cel) (Experimental)
  Interventions: Biological: Obecabtagene autoleucel (obe-cel)

INTERVENTIONS:
Biological: Obecabtagene autoleucel (obe-cel) — Obecabtagene autoleucel (obe-cel) given as a single infusion.

SUMMARY:
The main purpose of this study is to evaluate if obe-cel is safe or causes any side effects in adults with refractory progressive MS. The study also plans to assess if obe-cel can show early signs of efficacy in MS. The trial includes only 1 group of patients (single-arm). The study population comprises patients with progressive forms of MS, not responsive to highly effective therapies.

Upon confirmation of study eligibility, patients will receive fludarabine and cyclophosphamide (types of chemotherapy, used here for lymphodepletion) over 1 to 3 days in preparation for receiving a single obe-cel infusion.

Patients will be checked closely in the 28 days following obe-cel treatment. After this, patients will be monitored to evaluate safety and efficacy up to 24 months.

DETAILED DESCRIPTION:
This is a Phase 1 study to determine the safety, tolerability, and preliminary efficacy of obe-cel in participants with refractory progressive forms of multiple sclerosis.

The study comprises 3 periods:

Screening Period: From Day -30 to enrolment Treatment Period: From day of enrolment to End of Treatment (EOT) or Day 1 - Patients will be evaluated to confirm eligibility for lymphodepletion, and thereafter receive lymphodepletion to enhance treatment efficacy and CD19 chimeric antigen receptor (CAR) T cell survival.

Obe-cel Administration: If the participant's eligibility for receiving obe-cel infusion is confirmed, the participant is to receive a single obe cel infusion on Day 1.

Post treatment Period: From Day 1 to End of Study all participants will be followed up for efficacy and safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent for participation in the study.
* Ability and willingness to adhere to the protocol's Schedule of Activities and other requirements.
* Participants must be 18 to 60 years of age inclusive at the time of signing the informed consent form.
* A female participant is eligible to participate if she is not pregnant or breastfeeding.
* Current diagnosis of PMS.
* Must have been treated previously with 2 disease-modifying therapies

Exclusion Criteria:

* Any medications prohibited by the protocol.
* Highly active multiple sclerosis.
* Diagnosis of another autoimmune central nervous system condition.
* Active or uncontrolled fungal, bacterial, viral infection.
* History of malignant neoplasms unless disease-free for at least 24 months.
* History of heart, lung, kidney, liver transplant or hematopoietic stem cell transplant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2029-08-15 (Estimated); Study Completion 2029-08-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the tolerability of obe cel in participants with refractory forms of progressive multiple sclerosis (PMS) | Up to Day 28
  Percentage of participants receiving obe-cel who experience dose-limiting toxicities
To evaluate the safety of obe-cel in participants with refractory forms of progressive multiple sclerosis (PMS) | Up to end of study
  To evaluate the safety of obe-cel in participants with refractory forms of progressive multiple sclerosis (PMS)

SECONDARY OUTCOMES:
To evaluate the preliminary efficacy of obe-cel in participants with refractory forms of PMS using Expanded Disability Status Scale (EDSS) - Change from baseline in EDSS | Up to Month 24
  The EDSS is based on a standardized neurological examination focussing on assessment of 7 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel / bladder and cerebral). The range of the EDSS includes 20 half steps from 0 to 10, with EDSS step 0 corresponding to a completely normal examination and EDSS step 10 to death due to MS.
To evaluate the preliminary efficacy of obe-cel in participants with refractory forms of PMS using Timed 25-foot Walk Test (T25FWT). | Up to Month 24
  Change from baseline in T25FWT
To evaluate the preliminary efficacy of obe-cel in participants with refractory forms of PMS using 9-hole Peg Test (9-HPT) | Up to Month 24
  Change from baseline in 9-HPT
To evaluate the preliminary efficacy of obe-cel in participants with refractory forms of PMS using Symbol Digit Modalities Test (SDMT) | Up to Month 24
  Change from baseline in SDMT

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospital (UCLH), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No